CLINICAL TRIAL: NCT05603507
Title: Inspiratory Muscle Training Effects on Pulmonary Function and Quality of Life in Children With Chest Burn
Brief Title: Inspiratory Muscle Training in Children With Chest Burn
Acronym: chestburn
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qassim University (Other)
Collaborators: Cairo University (Other); Prince Sattam Bin Abdulaziz University (Other)
Responsible Party: Principal Investigator, Maged Basha, Assistant Professor, College of Medical Rehabilitation, Qassim University, Qassim University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RHPT/0020/0082
Record Dates: First submitted 2022-10-26; First posted 2022-11-02 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Burns; Respiratory Function Impaired; Children
Keywords: chest burn; respiratory muscle strength; lung function
MeSH Terms: conditions — Burns; Respiratory Insufficiency | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- inspiratory muscle training group (Experimental): received both inspiratory muscle training and pulmonary rehabilitation
  Interventions: Other: inspiratory muscle training; Other: pulmonary rehabilitation
- pulmonary rehabilitation group (Sham Comparator): received only pulmonary rehabilitation and sham inspiratory muscle training
  Interventions: Other: pulmonary rehabilitation

INTERVENTIONS:
Other: inspiratory muscle training — training done with a pressure threshold-loading device
  Other Names: inspiratory resistance
  Arms: inspiratory muscle training group
Other: pulmonary rehabilitation — Circuit training of aerobic and resistive exercise
  Other Names: Aerobic and resistance training

SUMMARY:
8 weeks of inspiratory muscle training combined with a pulmonary rehabilitation program increases respiratory muscle strength, pulmonary function, functional capacity, and quality of life in chest burned children.

DETAILED DESCRIPTION:
The primary purpose of this study is to see how an inspiratory muscle training program along with a pulmonary rehabilitation program improved respiratory muscle strength, respiratory function and quality of life after children with chest burns were discharged from the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 10 to 18.
* Following hospital discharge.- Total body surface area (TBSA) of 30% to 50%.
* Chest burns.
* Deep partial to full thickness burns.
* Subjects who had a skin graft or who healed completely were also included.

Exclusion Criteria:

* - Participants who had a nonhealing or open wound.
* Congenital diaphragmatic hernia.
* Chest wall deformity.
* Cardiac or pulmonary problems.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2022-04-09 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
maximal inspiratory pressure | 1 week after hospital discharge
  performed using an electronic respiratory pressure meter
maximal inspiratory pressure | 8 weeks
  performed using an electronic respiratory pressure meter
maximal expiratory pressure | 1 week after hospital discharge
  performed using an electronic respiratory pressure meter
maximal expiratory pressure | 8 weeks
  performed using an electronic respiratory pressure meter
Pulmonary function test, forced expiratory volume in the first second | 1 week after hospital discharge
  performed using a spirometer, the FEV1 (forced expiratory volume in the first second) was recorded.
Pulmonary function test, forced expiratory volume in the first second | 8 weeks
  performed using a spirometer, the FEV1 (forced expiratory volume in the first second) was recorded.
Pulmonary function test, forced vital capacity | 1 week after hospital discharge
  performed using a spirometer, the FVC (forced vital capacity) was recorded.
Pulmonary function test, forced vital capacity | 8 weeks
  performed using a spirometer, the FVC (forced vital capacity) was recorded.
Pulmonary function test, FEV1/FVC ratio | 1 week after hospital discharge
  performed using a spirometer, (forced expiratory volume in the first second/ forced vital capacity) FEV1/FVC ratio was recorded.
Pulmonary function test, FEV1/FVC ratio | 8 weeks
  performed using a spirometer, (forced expiratory volume in the first second/ forced vital capacity) FEV1/FVC ratio was recorded.

SECONDARY OUTCOMES:
Functional exercise capacity | 1 week after hospital discharge
  assessed using the six-minute walk test
Functional exercise capacity | 8 weeks
  assessed using the six-minute walk test
Health related Quality of Life | 1 week after hospital discharge
  assessed using the validated cross-culturally adapted version of the Pediatric Quality of life, The Peds-QL is a 23-item scale. Participants scored on a 5-point Likert scale ranging from 0 (never an issue) to 4 (almost always a problem). Following that, the item scores are decoded and linearly transformed to a 100-point scale. The psychosocial functioning summary score and physical functioning summary score were used for this study. A score of 100 indicates the highest functional status, while a score of 0 indicates the lowest functional status.
Health related Quality of Life | 8 weeks
  assessed using the validated cross-culturally adapted version of the Pediatric Quality of life, The Peds-QL is a 23-item scale. Participants scored on a 5-point Likert scale ranging from 0 (never an issue) to 4 (almost always a problem). Following that, the item scores are decoded and linearly transformed to a 100-point scale. The psychosocial functioning summary score and physical functioning summary score were used for this study. A score of 100 indicates the highest functional status, while a score of 0 indicates the lowest functional status.

CONTACTS AND LOCATIONS:
Overall Officials: Ragab Elnaggar, PhD, Study Chair — Prince Sattam Bin Abdulaziz University; Alshimaa Azab, PhD, Study Director — Prince Sattam Bin Abdulaziz University
Locations (1):
- Outpatient Clinic of College of Applied Medical Sciences, Prince Sattam bin Abdulaziz University, Al Kharj, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
The data sets generated during and/or analyzed during the current study are available from the corresponding author on reasonable request.
Supporting Information: Study Protocol, ICF
Time Frame: 6 months after publication
Access Criteria: relevance to the topic of the study and approval of all co-authors within 1 month of receiving the request.

REFERENCES:
- [Background] Willis CE, Grisbrook TL, Elliott CM, Wood FM, Wallman KE, Reid SL. Pulmonary function, exercise capacity and physical activity participation in adults following burn. Burns. 2011 Dec;37(8):1326-33. doi: 10.1016/j.burns.2011.03.016. Epub 2011 May 6. PMID 21530086
- [Result] Laszlo G. Standardisation of lung function testing: helpful guidance from the ATS/ERS Task Force. Thorax. 2006 Sep;61(9):744-6. doi: 10.1136/thx.2006.061648. PMID 16936234